CLINICAL TRIAL: NCT02333500
Title: Pilot Study: a Comparative Study Between Serum Levels of Oxytocin and Incitement to Use Olfactory Stimuli in Restrictive Anorexia Nervosa in Adolescents
Brief Title: Oxytocin and Incitement to Use Olfactory Stimuli in Restrictive Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-AOI-06
Record Dates: First submitted 2014-12-26; First posted 2015-01-07 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2018-07

CONDITIONS: Anorexia
MeSH Terms: conditions — Anorexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- olfactory workshop (Experimental): Influence of sensory therapy on the rate of oxytocin
  Interventions: Other: olfactory workshop
- other workshop (Active Comparator): Influence of other workshop on the rate of oxytocin
  Interventions: Other: other workshop
- control group (Other): Rate of oxytocin of the control group
  Interventions: Other: No intervention

INTERVENTIONS:
Other: olfactory workshop — olfactory workshop
  Arms: olfactory workshop
Other: other workshop — other workshop: discussion group, dance and body Expression
  Arms: other workshop
Other: No intervention — control group
  Arms: control group

SUMMARY:
This prospective pilot study will compare adolescents with restrictive anorexia nervosa who participated for 3 months at olfactory workshops, patients who did not, and healthy patients.The groups will be evaluated before the workshops and after three months, with the wanting score after olfactory stimuli and with serum oxytocin level.

DETAILED DESCRIPTION:
The restrictive anorexia nervosa (AN) in adolescents is an eating disorder with decreased desire to eat (wanting) following olfactory stimulation. Oxytocin is an hormone involved in the neuromodulation of eating behavior, but also involved in olfactory perception in schizophrenia patients, and in social cognition in patients with autism. Its plasma level was found low in anorexic patients compared to control subjects.

Because of the similarity in disorders of social cognition between these three diseases, we assume that the desire to eat evoked by olfactory perception varies with the plasma oxytocin levels.

With a prospective pilot study we will compare patients with AN who participated for 3 months at olfactory workshops, AN patients who did not, and healthy patients.

The groups will be evaluated before the workshops and after three months, with the wanting score after olfactory stimuli and with serum oxytocin level.

One application of this study will be the use of ocytocyne nasal spray to increase the eating desire and to allow weight regain

ELIGIBILITY:
Inclusion Criteria:

* Medical-Review
* Female or male -Sexe,
* 11 to 18 years
* Anorexia nervosa diagnosed according to the criteria DSM V
* Outpatient care or hospitalization
* Be able to answer the clinicals evaluations questionnaires
* Affiliated to social security
* Consentement of the legal representative and the patient

Exclusion Criteria:

* Somatic comorbidity associated with diabetes, celiac disease, brain tumor
* Intolerance odors, predisposed to develop asthma and / or respiratory allergies Pathologie chronic rhino-sinus
* Hyposmiques or anosmic
* Patients not of an inclusion criteria

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Score "Wanting" to olfactory stimuli | at 3 months

SECONDARY OUTCOMES:
Oxytocin serum level | at 3 months
Body mass index | at 3 months
Scores to clinical scales | at 3 months
Scores to hedonicity scale | at 3 months
Scores to "liking"-"wanting" tests | at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Florence ASKENAZY, PU-PH, Principal Investigator — Hôpitaux pediatriques CHU de Nice Fondation Lenval
Locations (1):
- Fondation Lenval Hôpitaux pediatriques CHU de Nice Fondation Lenval, Nice, France